CLINICAL TRIAL: NCT04453605
Title: Determining All Cause Morality and Cardiovascular Mortality Risk in Individuals With Neo-diagnosed Type 2 Diabetes
Brief Title: Phenotyping Individuals With Neo-diagnosed Type 2 Diabetes at Risk for All-cause Mortality
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Anna Solini, Associate Professor, University of Pisa
Other Study IDs: AS0006
Record Dates: First submitted 2020-05-07; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes; Vascular Diseases; Cardiac Disease
Keywords: neo-diagnosed type 2 diabetes; all-cause mortality; cardiovascular mortality
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with neo-diagnosed type 2 diabetes: Patients referring for the first time to the outpatient diabetes clinic in the department of Internal Medicine between January 2008 and December 2015 and matching the inclusion criteria.
  Interventions: Other: standard treatments

INTERVENTIONS:
Other: standard treatments — patients were treated according to the good clinical practice recommended by the international guidelines, and followed a six-month or an yearly calendar of follow-up visits

SUMMARY:
Prevalence of type 2 diabetes (T2D) is increasing worldwide over the last two decades; in these patients the rate of all-cause and cardiovascular (CV) mortality is several folds higher than in the general population, configuring a major public health problem. The clinical phenotype is the main determinant of such high mortality risk; however, a relevant role is played by the disease duration, with a significant interaction with metabolic control. However, for T2D the diagnosis does not correspond to the true onset of the disease, and a high lethality rate also in patients with recent onset of the disease cannot be excluded. Robust evidence supports this hypothesis, showing as in subjects with new-onset T2D, the mortality risk is superimposable, and even higher, than that observed in people with overt and long-term T2D. In this complex scenario, it would be desirable an early identification of high-risk patients, in which an accurate estimation of risk of complications, coupled with appropriate and timely interventions, might help in reducing the risk of encountering premature mortality. The present study was design to address this specific issue.

DETAILED DESCRIPTION:
Patients referring for the first time to the outpatient diabetes clinic in the department of Internal Medicine between January 2008 and December 2015 and matching the inclusion criteria were recruited.

Diagnosis was confirmed on the basis of the Oral Glucose Tolerance Test (OGTT) or HbA1c ≥6.5% plus fasting blood glucose ≥126 mg/dl.

Anthropometric measurements were recorded, arterial pressure and vital parameters were registered, and blood samples were collected for routine analyses. Complete blood count, glucose, HbA1c, Serum Glutamic Oxaloacetic Transaminase (sGOT), Serum Glutamic Pyruvic Transaminase (sGPT), uric acid, were determined by standard techniques. Total and HDL cholesterol and triglycerides were assayed through the automated spectrophotometer, enzymatic colorimetric method, COBAS INTEGRA using commercial kits (Roche Diagnostics). Serum creatinine was measured by Jaffe' method, and estimated glomerular filtration rate (eGFR) was calculated according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.

Previous major acute CV events, including myocardial infarction, stroke, foot ulcer/gangrene/amputation and coronary, carotid and lower limb revascularisation, were adjudicated based on hospital discharge records.

At the end of the baseline visit, patients were treated according to the good clinical practice recommended by the international guidelines, and followed a six-month or an yearly calendar of follow-up visits, until death or until 31 December 2018. All-cause mortality was assessed by checking the vital status of study participants on 31 December 2018; to this aim, investigators interrogated the Italian Health Card database, which provides updated information on all current Italian residents.

Incident major acute cardiovascular events were registered on the basis of clinical records every year; retinopathy onset was assessed by fundoscopy on a yearly basis.

ELIGIBILITY:
Inclusion Criteria:

* age ≥30 years
* personal history of known T2D lasting not more than six months
* diagnosis confirmed on the basis of the OGTT or HbA1c ≥6.5% plus fasting blood glucose ≥126 mg/dl

Exclusion Criteria:

* longstanding disease duration
* type 1 diabetes
* diabetes secondary to steroid therapy
* active cancer

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referring for the first time to the outpatient diabetes clinic in the department of Internal Medicine between January 2008 and December 2015 and matching the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who died during the study | At 31 December 2018
  The number of participants who died during the study was assessed by checking the vital status of study participants on 31 December 2018; to this aim, we interrogated the Italian Health Card database, which provides updated information on all current Italian residents.
Incidence of cardiovascular disease | At 31 December 2018
  Incident major acute cardiovascular events were registered on the basis of clinical records every year
Incidence of microvascular complication | At 31 December 2018
  Retinopathy onset was assessed by fundoscopy on a yearly basis.

SECONDARY OUTCOMES:
Change of renal function through study completion (an average of 5 year) | From baseline until the end of observation or the date of death from any cause, whichever came first, assessed up to 60 months.
  Serum creatinine was measured by Jaffe' method and expressed by mg/dl. It was used to calculate eGFR according to the CKD-EPI formula.
Change of blood glucose through study completion (an average of 5 year) | From baseline until the end of observation or the date of death from any cause, whichever came first, assessed up to 60 months.
  Blood glucose was expressed in mg/dl and was determined by standard techniques.
Change of HbA1c through study completion (an average of 5 year) | From baseline until the end of observation or the date of death from any cause, whichever came first, assessed up to 60 months.
  HbA1c was expressed as percentage or mmol/l and was determined by standard techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Solini, MD, PhD, Principal Investigator — University of Pisa
Locations (1):
- University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whiting DR, Guariguata L, Weil C, Shaw J. IDF diabetes atlas: global estimates of the prevalence of diabetes for 2011 and 2030. Diabetes Res Clin Pract. 2011 Dec;94(3):311-21. doi: 10.1016/j.diabres.2011.10.029. Epub 2011 Nov 12. PMID 22079683
- [Background] Tancredi M, Rosengren A, Svensson AM, Kosiborod M, Pivodic A, Gudbjornsdottir S, Wedel H, Clements M, Dahlqvist S, Lind M. Excess Mortality among Persons with Type 2 Diabetes. N Engl J Med. 2015 Oct 29;373(18):1720-32. doi: 10.1056/NEJMoa1504347. PMID 26510021
- [Background] Gregg EW, Zhuo X, Cheng YJ, Albright AL, Narayan KM, Thompson TJ. Trends in lifetime risk and years of life lost due to diabetes in the USA, 1985-2011: a modelling study. Lancet Diabetes Endocrinol. 2014 Nov;2(11):867-74. doi: 10.1016/S2213-8587(14)70161-5. Epub 2014 Aug 12. PMID 25128274
- [Background] Ghouse J, Isaksen JL, Skov MW, Lind B, Svendsen JH, Kanters JK, Olesen MS, Holst AG, Nielsen JB. Effect of diabetes duration on the relationship between glycaemic control and risk of death in older adults with type 2 diabetes. Diabetes Obes Metab. 2020 Feb;22(2):231-242. doi: 10.1111/dom.13891. Epub 2019 Nov 18. PMID 31596048
- [Background] Gimeno Orna JA, Blasco Lamarca Y, Campos Gutierrez B, Molinero Herguedas E, Lou Arnal LM. [Morbidity and mortality cardiovascular risk in dependence of type 2 diabetes duration]. Clin Investig Arterioscler. 2014 May-Jun;26(3):122-30. doi: 10.1016/j.arteri.2013.11.010. Epub 2014 Jan 23. Spanish. PMID 24461345
- [Background] Herrington WG, Alegre-Diaz J, Wade R, Gnatiuc L, Ramirez-Reyes R, Hill M, Solano-Sanchez M, Baigent C, Lewington S, Collins R, Tapia-Conyer R, Peto R, Kuri-Morales P, Emberson JR. Effect of diabetes duration and glycaemic control on 14-year cause-specific mortality in Mexican adults: a blood-based prospective cohort study. Lancet Diabetes Endocrinol. 2018 Jun;6(6):455-463. doi: 10.1016/S2213-8587(18)30050-0. Epub 2018 Mar 19. PMID 29567074
- [Background] Huo L, Magliano DJ, Ranciere F, Harding JL, Nanayakkara N, Shaw JE, Carstensen B. Impact of age at diagnosis and duration of type 2 diabetes on mortality in Australia 1997-2011. Diabetologia. 2018 May;61(5):1055-1063. doi: 10.1007/s00125-018-4544-z. Epub 2018 Feb 22. PMID 29473119
- [Background] Huang Y, Cai X, Mai W, Li M, Hu Y. Association between prediabetes and risk of cardiovascular disease and all cause mortality: systematic review and meta-analysis. BMJ. 2016 Nov 23;355:i5953. doi: 10.1136/bmj.i5953. PMID 27881363
- [Background] Smith NL, Barzilay JI, Kronmal R, Lumley T, Enquobahrie D, Psaty BM. New-onset diabetes and risk of all-cause and cardiovascular mortality: the Cardiovascular Health Study. Diabetes Care. 2006 Sep;29(9):2012-7. doi: 10.2337/dc06-0574. PMID 16936145